CLINICAL TRIAL: NCT06077019
Title: Role of Lung Function, Airway Inflammation and Bronchial Hyper Reactivity for Exercise Capacity in Well-trained Individuals
Brief Title: Role of Lung Function for Exercise Capacity in Well-trained Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morten Hostrup, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CHRON_INDAC_VIL
Record Dates: First submitted 2023-09-20; First posted 2023-10-11 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Exercise Performance
MeSH Terms: interventions — vilanterol; fluticasone furoate; indacaterol; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vilanterol (Experimental): Participants inhale vilanterol + fluticasone furoat
  Interventions: Drug: Vilanterol and Fluticasone Furoate
- Indacaterol (Experimental): Participants inhale indacaterol + mometasone furoate
  Interventions: Drug: Indacaterol and Mometasone Furoate
- Placebo (Placebo Comparator): Participants inhale placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vilanterol and Fluticasone Furoate — Participants inhale 25 µg vilanterol + fluticasone furoate daily
  Arms: Vilanterol
Drug: Indacaterol and Mometasone Furoate — Participants inhale 125 µg indacaterol + mometasone furoate daily
  Arms: Indacaterol
Drug: Placebo — Participants inhale placebo daily
  Arms: Placebo

SUMMARY:
The purpose of the project is to investigate exercise performance in humans following prolonged inhalation of beta2-agonists vilanterol + fluticasone furoate or indacaterol + mometasone furoate

ELIGIBILITY:
Inclusion Criteria:

* Age 18-39
* Physically active > 5 h weekly
* Maximal oxygen consumption classified as high or very high

Exclusion Criteria:

* Diagnosed with severe asthma and been in treatment with long-acting beta2-agonist/corticosteroid
* ECG abnormality
* ACQ score > 1.5
* Severe bronchial hyperreactivity as determined by mannitol test
* FEV1/FVC ratio < 0.7 determined with spirometry
* Chronic illness determined to be a potential risk for participant during study
* In chronic treatment with medication that may interfere with study results
* Pregnancy
* Smoker
* Blood donation during the past 3 months

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity during a time trial | Through study completion, an average of 8 weeks
  Mean power output measured in Watts during a time trial on a bike ergometer

SECONDARY OUTCOMES:
Lung function | Through study completion, an average of 8 weeks
  Forced expiratory volume in 1 second (FEV1) measured by spirometry before and after time trial with and without beta2-agonist induced bronchodilation

OTHER OUTCOMES:
Airway inflammation | Through study completion, an average of 8 weeks
  Measured by fractional nitric oxide in expired air
Mannitol induced bronchial hyper reactivity | Through study completion, an average of 8 weeks
  Assessed by decreases in FEV1 as dose response to cumulative doses of mannitol
Exercise induced bronchial hyper reactivity | Through study completion, an average of 8 weeks
  Assessed by decreases in FEV1 after maximal exercise
Quadriceps muscle strength | Through study completion, an average of 8 weeks
  Assessed by maximal isometric contraction torque
Lean body mass | Through study completion, an average of 8 weeks
  Measured with DXA-scanning
Fat mass | Through study completion, an average of 8 weeks
  Measured with DXA-scanning

CONTACTS AND LOCATIONS:
Overall Officials: Morten Hostrup, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data set will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Deidentified data set will be shared upon reasonable request.